CLINICAL TRIAL: NCT03230578
Title: Perspectives on Prescribing Hormonal Contraception Among Rural New Mexicans
Acronym: PHARM
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Eve Espey, Chair of OB/GYN, University of New Mexico
Other Study IDs: 17-237
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Contraception
Keywords: Pharmacists; Prescriptions
MeSH Terms: interventions — Pharmacists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacists: Actively employed and currently licensed and working in rural counties in New Mexico.
  Interventions: Other: Pharmacists & women's perspectives on pharmacist prescribed hormonal contraception
- Women: Reproductive age, 18-45 years old from rural counties in New Mexico and who are fluent in English.
  Interventions: Other: Pharmacists & women's perspectives on pharmacist prescribed hormonal contraception

INTERVENTIONS:
Other: Pharmacists & women's perspectives on pharmacist prescribed hormonal contraception — The goal of this study is to identify the thoughts and perceptions of pharmacy access to hormonal contraception among rural women and pharmacists. This will be key in order to address concerns or perceived barriers in order to inform the implementation of this program.

SUMMARY:
The goal of this study is to identify the thoughts and perceptions of pharmacy access to hormonal contraception among rural women and pharmacists. This will be key in order to address concerns or perceived barriers in order to inform the implementation of this program.

DETAILED DESCRIPTION:
There are no studies examining New Mexico pharmacists' interest in prescribing hormonal contraceptives or rural New Mexican women's support for pharmacist prescribed hormonal contraceptives. However, some states where pharmacists already prescribe contraception have experienced difficulties in implementing the education, infrastructure, and financial support necessary to provide hormonal contraception in the community pharmacy setting. Nationwide, 68% of women reported that they would utilize pharmacist prescribed hormonal contraception and cited benefits such as convenient hours and locations of pharmacies. The goal of this study is to identify the thoughts and perceptions of pharmacy access to hormonal contraception among rural women and pharmacists. This will be key in order to address concerns or perceived barriers in order to inform the implementation of this program.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacists: actively employed and currently licensed and working in rural counties in New Mexico.
* Women: Reproductive age, 18-45 years old from rural counties in New Mexico and who are fluent in English.

Exclusion Criteria:

* Pharmacists: decline to participate or work outside the defined rural areas, not currently employed or licensed.
* Women: younger than 18 or older than 45, living in urban areas (Albuquerque and Las Cruces).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our study is qualitative and not meant to capture a representative sample of the state's population, but rather capture a diverse array of opinions regarding hormonal contraception.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Pharmacist interview objective | 8/1/17-7/16/18
  To explore pharmacist perspectives on providing prescriptions for hormonal contraceptives, specifically identifying perceived barriers and facilitators to implementation.
Women interview objective | 8/1/17-7/16/18
  1.2. To explore women's perspectives on receiving hormonal contraception prescribed by pharmacists.
Hypothesis to be tested | 8/1/17-7/16/18
  Rural women and pharmacists across New Mexico will be supportive of prescriptive authority and pharmacy access to hormonal contraceptives.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Espey, MD, Principal Investigator — University of New Mexico, OB/GYN
Locations (1):
- Eve Espey, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Herman A, McCauley G, Thaxton L, Borrego M, Sussman AL, Espey E. Perspectives on prescribing hormonal contraception among rural New Mexican pharmacists. J Am Pharm Assoc (2003). 2020 Sep-Oct;60(5):e57-e63. doi: 10.1016/j.japh.2020.02.026. Epub 2020 Apr 2. PMID 32249171